CLINICAL TRIAL: NCT04393311
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study of the Safety and Efficacy of Ulinastatin for the Treatment of COVID-19 in Hospitalized Patients
Brief Title: Ulinastatin for the Treatment of COVID-19 in Hospitalized Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinuation of drug candidates
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56639
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ulinastatin (Experimental): Patients will receive ulinastatin via IV infusion every 8 hours for up to 5 days or until hospital discharge (whichever is earlier).
  Interventions: Drug: Ulinastatin
- Placebo (Placebo Comparator): Patients will receive placebo to match ulinastatin via IV infusion every 8 hours for up to 5 days or until hospital discharge (whichever is earlier).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ulinastatin — Ulinastatin administered via IV infusion (200,000/infusion)
  Arms: Ulinastatin
Drug: Placebo — Placebo to match ulinastatin administered via IV infusion
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of intravenous (IV) infusion of ulinastatin compared to placebo with respect to time to recovery, disease severity, need for ventilator support, and mortality in patients with COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Signs and symptoms suggestive of COVID-19 infection
* Laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection ≤7 days before randomization
* Currently hospitalized or in an emergency department with planned hospitalization
* Peripheral capillary oxygen saturation (SpO2) <93% on room air at Screening

Exclusion Criteria:

* Simultaneous participation in any other clinical study incompatible with this one
* Treatment with an antibody immunotherapy within 4 weeks of Screening
* Requirement for mechanical ventilation or ECMO at Screening
* Hypotension at Screening
* Severe liver injury defined as AST or ALT ≥5x the upper limit of normal
* Severe kidney failure defined as an estimated glomerular filtration rate (eGFR) <30 mL/min
* Pregnancy or breastfeeding
* > 120 hours between admission and signing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | Up to 29 days
  Time to recovery, defined as attaining a score of 6, 7, or 8 on the COVID-19 disease severity scale, an 8 point ordinal scale used in the NIH Adaptive COVID-19 Treatment Trial (ACTT; NCT04280705).
  1. = Death;
  2. = Hospitalized and on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  3. = Hospitalized and on non-invasive ventilation or high-flow oxygen devices;
  4. = Hospitalized and requiring supplemental oxygen;
  5. = Hospitalized and not requiring supplemental oxygen but requiring ongoing medical care (COVID-19-related or otherwise);
  6. = Hospitalized and not requiring supplemental oxygen and no longer requiring ongoing medical care;
  7. = Not hospitalized, limitation on activities and/or requiring home oxygen;
  8. = Not hospitalized, no limitation on activities

SECONDARY OUTCOMES:
COVID-19 disease severity scale score on Day 8 | Day 8
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
COVID-19 disease severity scale score on Day 15 | Day 15
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
COVID-19 disease severity scale score on Day 22 | Day 22
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
COVID-19 disease severity scale score on Day 29 | Day 29
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
Incidence of mortality at Day 29 | 29 days
Incidence of in-hospital mortality | Up to 29 days
Number of days alive and not on mechanical ventilator or ECMO in the 28 days following first dose | Up to 29 days
Number of patients with resolution of symptoms defined as score of 8 on the 8-point ordinal scale at Day 29 | Day 29
Number of patients alive and free of respiratory failure defined as score of 4, 5, 6, 7, or 8 on the 8-point ordinal scale at Day 29 | Day 29
Duration of mechanical ventilation | Up to 29 days
  For patients requiring mechanical ventilation.
Duration of ECMO | Up to 29 days
  For patients requiring mechanical ECMO.
Duration of noninvasive ventilation | Up to 29 days
  For patients requiring non-invasive ventilation
Duration of ICU stay | Up to 29 days
  For patients admitted to ICU
Duration of hospital stay | Up to 29 days
Change in oxygen saturation | Between screening and 24 hours after last dose (up to 6 days)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin V Grimes, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.